CLINICAL TRIAL: NCT02619097
Title: Safety & Pharmacokinetics of Pegolsihematide for Treatment of Anemia Patient With Myelodysplastic Syndromes
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-EPOP1b
Record Dates: First submitted 2015-11-20; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Myelodysplastic Syndromes; Anemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 0.08mg/kg (Experimental): Pegol-sihematide injection, 0.08mg/kg, single-dose
  Interventions: Drug: Pegol-sihematide injection
- 0.2mg/kg (Experimental): Pegol-sihematide injection, 0.2mg/kg, single-dose
  Interventions: Drug: Pegol-sihematide injection
- 0.33mg/kg (Experimental): Pegol-sihematide injection, 0.33mg/kg, single-dose
  Interventions: Drug: Pegol-sihematide injection
- 0.5mg/kg (Experimental): Pegol-sihematide injection, 0.5mg/kg, single-dose
  Interventions: Drug: Pegol-sihematide injection
- 0.7mg/kg (Experimental): Pegol-sihematide injection, 0.7mg/kg, single-dose
  Interventions: Drug: Pegol-sihematide injection

INTERVENTIONS:
Drug: Pegol-sihematide injection — single dose
  Other Names: EPO-018B

SUMMARY:
The primary objectives of the trial are to assess the safety and pharmacokinetics profile of pegolsihematide for treatment of anemia patient with myelodysplastic syndromes.

DETAILED DESCRIPTION:
The study started from the lowest dose, 0.08mg/kg, each group will enroll 4 to 6 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years, premenopausal women must have negative pregnancy test.
2. Documented diagnosis of myelodysplastic syndromes (MDS) according to World Health Organization (WHO) criteria, including refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), refractory cytopenia with multilineage dysplasia (RCMD), MDS-U, 5q-.
3. Meets International Prognostic Scoring System (IPSS) classification of low or intermediate-1 risk disease as determined by microscopic and standard cytogenetic analysis of the bone marrow during screening.
4. Never with erythropoietin agents treatment prior to enrollment.
5. Eastern cooperative oncology group (ECOG) performance status of 0 or 1 during screening.
6. Hemoglobin ≥7g/dL and ≤10g/dL, at least two detections during screening.
7. Adequate transferrin saturation (≥15%), ferritin (≥12ng/mL), folate (≥ lower limits of normal), vitamin B12 (≥ lower limits of normal)
8. Patients understand and are able to provide written informed consent.

Exclusion Criteria:

1. Pregnant or breast feeding women or women having positive pregnant test, women or men whose spouse plan to become pregnant with 4 weeks after the end of treatment .
2. Therapy-related or secondary MDS.
3. Previously diagnosed with intermediate-2 or high risk MDS per International Prognostic Scoring System (IPSS).
4. History of severe allergic or anaphylactic reactions or hypersensitivity to erythropoiesis-stimulating agents or polyethylene glycol.
5. History of red blood cell or blood transfusion during 4 weeks prior to enrollment.
6. Known other disease which can lead to anemia (including haemolytic disease and digestive tract hemorrhage).
7. Uncontrolled hypertension 2 weeks prior to enrollment, defined as systolic blood pressure ≥160mmHg or diastolic blood pressure ≥ 95mmHg.
8. Clinically significant systemic infection or uncontrolled chronic inflammatory disease (ie, rheumatoid arthritis, inflammatory bowel disease) as determined by the investigator at screening.
9. Evidence of bone marrow collagen fibrosis, biopsy argentaffin staining showed reticular fiber ≥＋＋.
10. History of deep venous thrombosis or arterial embolism within 12 months prior to enrollment.
11. History of cardiocerebrovascular events within 6 months prior to enrollment, include local ischemia, embolism, cerebral hemorrhage, transient ischemic attack, myocardial ischemia or other arterial thrombosis.
12. Any serious medical condition, lab abnormality or psychiatric illness within 6 months prior to enrollment.
13. History of malignancies other than curatively treated non-melanoma skin or in situ carcinoma.
14. Estimated survival time < 6 months.
15. Plan to get major surgery which will lead to massive bleeding during the study.
16. Treatment with any other investigational drug within 6 weeks prior to enrollment, or plan to participate in any other investigational drug during the study.
17. Any other condition not specifically noted above which, in the judgement of the investigator, would preclude the patient from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 28 days after injection
Maximum Plasma Concentration [Cmax] | 10min before injection to 336h after injection
Time to Maximum Plasma Concentration [Tmax] | 10min before injection to 336h after injection
Half-life [t1/2] | 10min before injection to 336h after injection
Area Under the Curve [AUC]). | 10min before injection to 336h after injection

SECONDARY OUTCOMES:
The changes of hemoglobin (g/L) after treatment | From date of recruitment until the date of biggest documented progression up to 28 weeks
The changes of reticulocyte (10^9/L) after treatment | From date of recruitment until the date of biggest documented progression up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Xiao, Doctor, Study Chair — Hospital of Blood Diseases, Chinese Academy of Medical Sciences
Locations (1):
- Hospital of Blood Diseases, Chinese Academy of Medical Sciences, Tianjin, China